CLINICAL TRIAL: NCT05156463
Title: Evaluating a Physical Activity Assessment and Counseling Index for Breast and Colon Cancer Survivors in Clinical Practice (The PAI Trial)
Brief Title: The PAI Trial for Breast and Colon Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Award not yet received and PI is transferring to a different institution
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Shirley Bluethmann, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00018917
Record Dates: First submitted 2021-11-16; First posted 2021-12-14 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Colon Cancer
Keywords: Adult Cancer Survivors; Geriatrics; Gerontology
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive standard follow-up survivorship care, an accelerometer to measure physical activity and NCCN (National Comprehensive Cancer Network) patient materials.
- Treatment (Experimental): Participants will receive same materials as standard of care group. In addition participants will use PAI Activity tool, Garmin activity tracker and exercise logs, and also receive periodic exercise coaching.
  Interventions: Combination Product: PAI Tool and Exercise Coaching

INTERVENTIONS:
Combination Product: PAI Tool and Exercise Coaching — Use of PAI tool and self-monitoring tools to increase physical activity and reduce sedentary behaviors. Participants will receive a personalized physical assessment and counseling from healthcare provider, exercise logs and a Garmin activity tracker to use between visits and 9 exercise coaching calls between clinical visits.
  Arms: Treatment

SUMMARY:
The purpose of the study is to determine if a Physical Activity Index (PAI) tool that collects measures on physical activity, strength training and sedentary behavior can be used in a clinical setting to monitor patient behavior and provide specific recommendations on how to achieve and maintain behavior goals. The tool will be used after treatment is completed in breast and colon cancer survivors and will test if physician counseling combined with patient self-monitoring improves physical activity and reduces sedentary behavior over time.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 60 years or older diagnosed with breast cancer and women or men ages 60 years or older diagnosed with colon cancer within the last 5 years
* ≥ 3 months post-completion of last prescribed treatment (i.e., Chemotherapy, radiation therapy or surgery)
* Stages I-III (no stage 0 or metastatic cases will be included)
* Able to understand spoken and written instructions in English
* Participate in 60 minutes or more of MVPA (moderate to vigorous-intensity physical activity)/week for previous 6 months
* Have internet access or access to data sharing plan
* Willing to come to four Penn State Health visits over the course of a year, completing requested questionnaires
* Willing to use Garmin Vivofit device, participate in exercise coaching sessions and complete exercise logs between visits

Exclusion Criteria:

* Prior respiratory, joint or cardiovascular problems precluding PA
* Metastatic disease
* Planned elective surgery during intervention/follow-up
* Exhibit gross cognitive impairment

We will not include any of the following vulnerable populations: adults unable to consent, individuals who are not yet adults, pregnant women, neonates, or prisoners.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer survivors Female/Male colon cancer survivors
Enrollment: 0 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Introduce PAI tool to increase PA and reduce sedentary behavior | 7 days prior to each visit clinical visit (Baseline, 3 months, 6 months, 12 months)
  PAI Tool: frequency and time spent in strenuous moderate and mild PA over 7 days and self reported television time or sedentary screen time per week
Change in activity as measured by Community Healthy Activities Model Program for Seniors (CHAMPS) Questionnaire for Older Adults | Baseline, 3 months, 6 months,12 months
  This self-report questionnaire assesses weekly frequency and duration of a variety of lifestyle physical activities that are meaningful and appropriate for older adults. Scores are recorded based on number of repetitions the activity was completed and the hours spent doing the activity from less than 1 hour to 9 or more hours.
Use of Actigraph to measure changes in activity and sedentary behavior | 7 days prior to each clinical visit (Baseline, 3 months, 6 months, 12 months)
  Activity patterns and sedentary behavior based on 7 days of wear before clinical visit

SECONDARY OUTCOMES:
Modified Cancer and Aging Research Group (CARG) plus National Health and Nutrition Examination Survey (NHANES) and Patient-Reported Outcomes Measurement Information System (PROMIS) Geriatric Assessment Study Patient Questionnaire | Baseline, 3 months, 6 months,12 months
  Aggregated assessment of self-reported information about demographic data, daily activities, nutritional status, medication use and health behaviors.
Exercise Self-Efficacy Scale This scale assesses an individual's beliefs in their ability to continue exercising on a 3 time/week basis at moderate intensities for 40+ min. per session in the future. | Baseline, 3 months, 6 months, 12 months
  For 8 items, participants indicate their confidence to execute the behavior on a 100-pt percentage scale comprised of 10-pt increments, ranging from 0% (not at all confident) to 100% (highly confident).

CONTACTS AND LOCATIONS:
Overall Officials: Shirley M Bluethmann, PhD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No